CLINICAL TRIAL: NCT04100330
Title: A Phase 2, Randomized, Open-Label, Multicenter Study of Ficlatuzumab in Combination With High-Dose Cytarabine (HiDAC) and HiDAC Alone in Adults With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study of Ficlatuzumab With HiDAC and HiDAC Alone in Adults With Relapsed or Refractory Acute Myeloid Leukemia
Acronym: CyFi2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Urgent shift among clinical sites toward efforts to combat COVID-19 pandemic;impacted feasibility of completing study within shelf-life of current IP supply
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-299-19-207
Record Dates: First submitted 2019-09-12; First posted 2019-09-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ficlatuzumab; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ficlatuzumab with HiDAC (Experimental): Ficlatuzumab 20 mg/kg intravenously (IV) on Days 1 and 15 in combination with cytarabine 2 g/m2 IV per day on Days 2 through 7. Up to two additional doses can be administered - on Day 29, or on Days 29 and 43, if prolonged myelosuppression is experienced.
  Interventions: Biological: Ficlatuzumab; Drug: Cytarabine
- HiDAC alone (Active Comparator): Cytarabine 2 g/m2 IV per day on Days 1 through 6
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Biological: Ficlatuzumab — Ficlatuzumab is a selective recombinant humanized hepatocyte growth factor (HGF) inhibitory immunoglobulin G subclass 1 monoclonal antibody which blocks the MET tyrosine kinase receptor.
  Other Names: AV-299
  Arms: Ficlatuzumab with HiDAC
Drug: Cytarabine — Cytarabine is a chemotherapy agent. Chemotherapy agents are medications that kill cancer cells.
  Other Names: Ara-C; Arabinosylcytosine

SUMMARY:
This is a Phase 2, randomized, open-label, multicenter study to evaluate the safety and efficacy of ficlatuzumab in combination with high-dose cytarabine (HiDAC) and HiDAC alone in subjects with relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML according to the WHO criteria, which defines relapsed or refractory to induction therapy as follows:

   1. First relapse within 12 months after date of first CR or CRi
   2. Persistent AML documented by bone marrow biopsy at least 29 days after Day 1 of the first induction cycle of cytotoxic chemotherapy
   3. Hypercellular bone marrow with greater than 20% cellularity and 10% blasts at least 14 days after the first induction cycle Day 1
2. Age ≥18 years
3. Prior induction therapy, consisting of no more than 2 cycles of cytotoxic chemotherapy with at least one of the cycles consisting of anthracycline and cytarabine with reasonable schedule/dose intensity according to the discretion of the Investigator
4. Histologically confirmed AML by hematopathology review performed within 4 weeks of study entry. Secondary AML due to progression of myelodysplastic syndrome or myeloproliferative neoplasms is acceptable for inclusion.
5. Prior treatment for myelodysplastic syndrome or myeloproliferative neoplasm with hypomethylating agent or targeted agent is acceptable for inclusion
6. Ejection fraction ≥40% by echocardiogram or multigated acquisition (MUGA) scan
7. Cytoreduction therapy with leukapheresis or hydroxyurea is allowed
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
9. Clinical laboratory values meeting the following criteria before Day 1 (Cycle 1, Day 1):

   1. An estimated glomerular filtration rate of ≥ 60mL/min based on Cockcroft-Gault equation calculated using serum creatinine levels
   2. Total bilirubin ≤2.0 mg/dL (≤3.0 mg/dL for subjects with known Gilbert's syndrome)
   3. Aspartate aminotransferase (AST) or ALT ≤2.5 × ULN, unless thought to be due to AML
   4. Activated partial thromboplastin time ≤1.5 × ULN and prothrombin time/international normalized ratio (PT/INR) ≤1.5 × ULN if not on anticoagulation therapy. Subjects receiving anticoagulation therapy with an agent such as warfarin or low-molecular weight heparin may be allowed to participate with the therapeutic range established before initiation of study treatment.
10. For female subjects of childbearing potential, documentation of negative serum pregnancy test before randomization
11. For female subjects of childbearing potential and male subjects whose sexual partners are of childbearing potential, agreement to use an effective method of contraception during the study and for at least 90 days after the last dose of ficlatuzumab. Effective birth control includes (a) intrauterine device plus 1 barrier method; (b) oral, implantable, or injectable contraceptive plus 1 barrier method; or (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).
12. Ability to give written informed consent and comply with protocol requirements

Exclusion Criteria:

1. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent or cytarabine
2. Acute promyelocytic leukemia (AML French-American-British classification M3)
3. More than 2 cycles of prior induction therapy for AML
4. Prior treatment with intermediate- or HiDAC (≥1 gm/m2)
5. Allogeneic or autologous hematopoietic cell transplantation within 90 days of study entry
6. Prior treatment with any other investigational drugs, biologics, or devices, within 4 weeks before Day 1
7. Active graft versus host disease or immunosuppression for prevention or treatment of graft versus host disease within 4 weeks of study entry
8. Chemotherapy or radiation therapy within 1 week before study entry, other than hypomethylating agents or hydroxyurea used for cytoreduction
9. Significant cardiovascular disease, including:

   1. Cardiac failure New York Heart Association class III or IV
   2. Myocardial infarction, severe or unstable angina within 6 months before Day 1
   3. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation)
10. Significant thrombotic or embolic events within 3 months before Day 1 (significant thrombotic or embolic events include, but are not limited to, venous thromboembolism, stroke, or transient ischemic attack). Catheter-related thrombosis is not a cause for exclusion. Diagnosis of deep vein thrombosis or pulmonary embolism is allowed if it occurred >3 months before Day 1 and anticoagulation therapy is completed before Day 1.
11. Any other medical condition or psychiatric condition that, in the opinion of the Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results
12. History of prior/concurrent malignancy whose natural history or ongoing treatment is expected to interfere with the safety or efficacy assessment of the intervention
13. Known seropositive or active HIV
14. Active hepatitis B or C infection
15. Uncontrolled systemic fungal, bacterial, or viral infections
16. For female subjects, pregnant or breastfeeding
17. Prior exposure to the investigational agent or anti-c-MET, or anti-HGF within 6 months before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 13 months (through study treatment completion)
  To estimate the overall response rate (ORR) (complete remission [CR] + CR with incomplete hematologic recovery [CRi]) of ficlatuzumab in combination with high-dose cytarabine (HiDAC) and HiDAC alone in adults with relapsed or refractory acute myeloid leukemia (AML)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Approximately 14 months (through 30 days after the last subject completes treatment)
  To evaluate the safety and tolerability of ficlatuzumab when administered with HiDAC and HiDAC alone
Overall Survival (OS) | For up to one year after the end of study treatment
  To estimate the overall survival (OS) rate of ficlatuzumab in combination with HiDAC and HiDAC alone in adults with relapsed or refractory AML
Disease-Free Survival (DFS) | For up to one year after the end of study treatment
  To estimate the disease-free survival (DFS) rate of ficlatuzumab in combination with HiDAC and HiDAC alone in subjects achieving CR

IPD SHARING:
Plan to Share IPD: No